CLINICAL TRIAL: NCT02337725
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of TVP-1012 at 1 mg in Early Parkinson's Disease Patients Not Treated With Levodopa
Brief Title: A Phase 3 Study of TVP-1012 (1 mg) in Early Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TVP-1012/CCT-001; U1111-1165-1302 (Registry Identifier: WHO); JapicCTI-152760 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TVP-1012 1 mg (Experimental): For 2 weeks during the run-in period, one tablet of placebo orally, once daily before or after breakfast, followed by 26 weeks during the treatment period, one tablet of TVP-1012 1 mg orally, once daily before or after breakfast.
  Interventions: Drug: TVP-1012
- Placebo (Placebo Comparator): For 2 weeks during the run-in period, one tablet of placebo orally, once daily before or after breakfast, followed by 26 weeks during the treatment period, one tablet of placebo orally, once daily before or after breakfast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TVP-1012 — TVP-1012 1mg Tablets
  Arms: TVP-1012 1 mg
Drug: Placebo — Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TVP-1012 (1 mg/day) administered to Japanese patients with early Parkinson's disease.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-group, phase 3 study to evaluate the efficacy and safety of TVP-1012 in Japanese participants with early Parkinson's disease.

The study period consisted of a 28-week trial period. The participants who fulfill the inclusion criteria and not meeting any of the exclusion criteria were enrolled, and randomized in a 1:1 ratio to either the 1 mg of TVP-1012 or the placebo group. In each treatment group, participants received either 1 mg of TVP-1012 or placebo once daily in a double-blinded manner.

ELIGIBILITY:
Inclusion Criteria:

Run-in period

* In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* The participant has a diagnosis of Parkinson's disease with at least two of the following signs: resting tremor, akinesia/bradykinesia, and muscle rigidity.
* The participant has a Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II + Part III total score of >=14 at the start of the run-in period.
* The participant has Modified Hoehn & Yahr stage 1 to 3 at the start of the run-in period.
* The participant has the Parkinson's disease diagnosed within 5 years prior to the start of the run-in period.
* The participant is an outpatient of either sex aged >= 30 and < 80 years.
* A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent to 1 month after the last dose of the investigational drug.

Treatment period

- The participant has a MDS-UPDRS Part II + Part III total score of >= 14 at baseline.

Exclusion Criteria:

Run-in period

* The participant has received any investigational medication within 90 days prior to the start of the run-in period.
* The participant has received TVP-1012 in the past.
* The participant is study site employee, an immediate family member, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
* Participant has donated 400 mL or more of his or her blood volume within 90 days prior to the start of the run-in period.
* The participant has unstable systemic disease.
* The participant has Mini-Mental State Examination (MMSE) score of <= 24 at the start of the run-in period.
* The participant has known or a history of schizophrenia, major or severe depression, or any other clinically significant psychiatric disease.
* The participant has a history of hypersensitivity or allergies to TVP-1012 (including any associated excipients) or selegiline.
* The participant has a history of clinically significant hypertension or other reactions associated with ingestion of tyramine-rich food (e.g., cheese, lever, herring, yeast, horsebean, banana, beer or wine).
* The participant has a history or concurrent of drug abuse or alcohol dependence.
* The participant has received neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, deep brain stimulation).
* The participant has received transcranial magnetic stimulation within 6 months prior to the start of the run-in period
* The participant has received amantadine or anticholinergic medication for >= 180 days.
* The participant has received selegiline, a levodopa-containing product or dopamine agonist for >= 90 days.
* The participant has received selegiline, pethidine, tramadol, reserpine or methyldopa within 90 days prior to the start of the run-in period.
* The participant has received a levodopa-containing product, dopamine agonist, amantadine or anticholinergic drug within 30 days prior to the start of the run-in period.
* The participant has received any psychoneurotic agent or antiemetic medication of dopamine antagonist within 14 days prior to the start of the run-in period. However, the participant has been receiving quetiapine or domperidone with a stable dose regimen for >= 14 days prior to the start of the run-in period may be included in the study.
* The participant has previously received a catechol-O-methyltransferase (COMT) inhibitor, droxidopa, zonisamide or istradefylline.
* The participant is required to take any of the prohibited concomitant medications or treatments.
* If female, the participant is pregnant or lactating or intending to become pregnant during this study, or within 1 month after the last dose of the investigational drug; or intending to donate ova during such time period.
* The participant has clinically significant neurologic, cardiovascular, pulmonary, hepatic (including mild cirrhosis), renal, metabolic, gastrointestinal, urological, endocrine, or hematological disease.
* The participant has clinically significant or unstable brain or cardiovascular disease, such as:

  * clinically significant arrhythmia or cardiac valvulopathy,
  * cardiac arrest of NYHA Class II or higher,
  * concurrent or a history of ischemic cardiac disease within 6 months prior to the start of the run-in period,
  * concurrent or a history of clinically significant cerebrovascular disease within 6 months prior to the start of the run-in period,
  * sever hypertension (systolic blood pressure of 180 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher),
  * clinically significant orthostatic hypotension (including those with systolic pressure decrease of 30 mmHg or more following postural change from supine/sitting position to standing position),
  * a history of syncope due to hypotension within 2 years prior to the start of the run-in period.
* The participant is required surgery or hospitalization for surgery during the study period
* Participant has a history of cancer within 5 years prior to the start of the run-in period, except cervix carcinoma in situ which has completely cured.
* The participant has acquired immunodeficiency syndrome (AIDS) [including human immunodeficiency virus (HIV) carrier], or hepatitis [including viral hepatitis carrier such as hepatitis B surface (HBs) antigen or hepatitis C antibody (HCV) positive]. However, the participant who has a negative result for HCV antigen or HCV-RNA can be included in the study.
* The participant who, in the opinion of the investigator or sub-investigator, is unsuitable for any other reason.

Treatment period

* The participant whose diagonosis of Parkinson's disease is ruled out by dopamine transporter scintigraphy performed during the run-in period if conducted.
* The participant has laboratory data meeting any of the following at the start of the run-in period:

  * Creatinine >= 2 x upper limit of normal (ULN)
  * Total bilirubin >= 2 x ULN
  * ALT or AST >= 1.5 x ULN
  * ALP >= 3 x ULN
* The participant has received any of the prohibited concomitant medications or treatments during the run-in period.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2015-02-07 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (55):
- Japan (55):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Touon, Ehime
  - Kitakyushu, Fukuoka
  - Onoshiro, Fukuoka
  - Asahikawa, Hokkaido
  - Iwamizawa, Hokkaido
  - Akashi, Hyōgo
  - Kobe, Hyōgo
  - Tsuchiura, Ibaragi
  - Tsukuba, Ibaragi
  - Morioka, Iwate
  - Takamatsu, Kagawa-ken
  - Fujisawa, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Gōshi, Kumamoto
  - Sendai, Miyagi
  - Matsumoto, Nagano
  - Higashisonogi-gun, Nagasaki
  - Nishisonogi-gun, Nagasaki
  - Tenri, Nara
  - Jouetsu, Niigata
  - Higashiosaka, Osaka
  - Suita, Osaka
  - Takatsuki, Osaka
  - Toyonaka, Osaka
  - Irima-gun, Saitama
  - Fuji, Shizuoka
  - Hamamatsu, Shizuoka
  - Izunokuni, Shizuoka
  - Shimono, Tochigi
  - Yoshinogawa, Tokushima
  - Bunkyo-ku, Tokyo
  - Fuchū, Tokyo
  - Kodaira, Tokyo
  - Meguro-ku, Tokyo
  - Nerima-ku, Tokyo
  - Ōta-ku, Tokyo
  - Setagaya-ku, Tokyo
  - Shibuya-ku, Tokyo
  - Akita
  - Aomori
  - Fukuoka
  - Fukushima
  - Hiroshima
  - Kochi
  - Kyoto
  - Niigata
  - Okayama
  - Osaka
  - Tokushima
  - Toyama
  - Wakayama
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hattori N, Takeda A, Takeda S, Nishimura A, Kitagawa T, Mochizuki H, Nagai M, Takahashi R. Rasagiline monotherapy in early Parkinson's disease: A phase 3, randomized study in Japan. Parkinsonism Relat Disord. 2019 Mar;60:146-152. doi: 10.1016/j.parkreldis.2018.08.024. Epub 2018 Sep 1. PMID 30205936

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 68 investigative sites in Japan, from 07-Feb-2015 to 15-Sep-2016.
Pre-assignment Details: Participants with diagnosis of Parkinson's disease were enrolled and received one tablet of placebo orally, once daily in a run-in period (Week -2 to 0). After that, the participants who fulfilled the inclusion criteria and did not meet any of the exclusion criteria at Week -2 and Week 0 were randomized in 1:1 to TVP-1012 1 mg or Placebo at Week 0.
Groups:
- TVP-1012 1mg: For 2 weeks during the run-in period, one tablet of placebo orally, once daily before or after breakfast, followed by 26 weeks during the treatment period, one tablet of TVP-1012 1 mg orally, once daily before or after breakfast.
Period: Overall Study
Arm/Group | Placebo | TVP-1012 1mg
Started | 126 | 118
Completed | 100 | 110
Not Completed | 26 | 8
Not completed — Pretreatment Event/AE before Treatment | 0 | 1
Not completed — Pretreatment Event/AE in Treatment | 8 | 3
Not completed — Major Protocol Deviation | 0 | 1
Not completed — Voluntary Withdrawal | 14 | 3
Not completed — Lack of Efficacy | 4 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set was defined as all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TVP-1012 1mg | Total
Number analyzed (Participants) | 126 | 118 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (8.81) | 67.4 (8.96) | 66.4 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 65 | 137
  Male | 54 | 53 | 107
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 126 | 118 | 244
Height [Mean (Standard Deviation); unit: cm] | 159.3 (9.24) | 158.8 (8.86) | 159.0 (9.04)
Weight [Mean (Standard Deviation); unit: kg] — Population: The number analyzed is the number of participants with data available for analysis.
  kg
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 56.97 (10.218) | 57.91 (11.803) | 57.42 (10.997)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2] Population: The number analyzed is the number of participants with data available for analysis.
  kg/m^2
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 22.35 (2.752) | 22.78 (3.303) | 22.56 (3.031)
Smoking Classification [Count of Participants; unit: Participants]
  Never Smoked | 75 | 64 | 139
  Current Smoker | 8 | 5 | 13
  Ex-Smoker | 43 | 49 | 92
Timing of Study Drug Dose [Count of Participants; unit: Participants]
  Before Breakfast | 60 | 59 | 119
  After Breakfast | 66 | 59 | 125
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: years] | 1.56 (1.237) | 1.97 (1.972) | 1.76 (1.644)
Modified Hoehn & Yahr Stage [Mean (Standard Deviation); unit: Units on a scale] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)).
  Units on a scale | 2.15 (0.615) | 2.18 (0.626) | 2.17 (0.619)
MDS-UPDRS Part II+III Total Score [Mean (Standard Deviation); unit: Scores on a scale] — Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part II+III Total Score was 0-188, with higher scores reflecting greater severity. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 33.8 (14.43) | 34.4 (16.95) | 34.1 (15.66)
MDS-UPDRS Part I Total Score [Mean (Standard Deviation); unit: Scores on a scale] — For MDS-UPDRS Part I (non-motor experiences of daily living) scores, the scale range for Part I Total Score was 0-52, with higher scores reflecting greater severity. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 5.7 (3.58) | 5.5 (3.83) | 5.6 (3.70)
MDS-UPDRS Part II Total Score [Mean (Standard Deviation); unit: Scores on a scale] — For MDS-UPDRS Part II (motor experiences of daily living) scores, the scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 7.0 (4.64) | 7.2 (5.47) | 7.1 (5.05)
MDS-UPDRS Part III Total Score [Mean (Standard Deviation); unit: Scores on a scale] — For MDS-UPDRS Part III (motor examination) scores, the scale range for Part III Total Score was 0-136, with higher scores reflecting greater severity. Population: The number analyzed is the number of participants with data available for analysis.
  Scores on a scale
    number analyzed (Participants) | 126 | 117 | 243
    (all) | 26.8 (11.59) | 27.2 (13.80) | 27.0 (12.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II + Part III Total Score
Description: Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retains the four-scale structure with a reorganization of the various subscale; (Part I; 13 items) non-motor experiences of daily living, (Part II; 13) motor experiences of daily living, (Part III; 34) motor examination, and (Part IV; 6) motor complications. Each items had 0-4 ratings, where 0 (normal) to 4 (severe) and score for each was summed to calculate the total scores. The scale range for Part II+III Total Score was 0-188, with higher scores reflecting greater severity.
Time Frame: From Baseline to Week 26 (LOCF)
Population: Full Analysis Set included all randomized participants who received at least 1 dose of the study drug for the treatment period. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 125 | 115
Units on a scale | 1.87 (0.752) | -4.52 (0.784)
Statistical Analysis 1: Comparison: Placebo vs TVP-1012 1mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -6.39, 95% CI 2-sided [-8.530 to -4.250] — Estimated Value was reported for the least squares mean difference between TVP-1012 1mg and Placebo (TVP-1012 1mg - Placebo)

2. Secondary Outcome: Change From Baseline in MDS-UPDRS Part I Total Score
Description: For MDS-UPDRS Part I (non-motor experiences of daily living) scores, the scale range for Part I Total Score was 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 125 | 116
Units on a scale | 0.98 (0.247) | 0.18 (0.257)

3. Secondary Outcome: Change From Baseline in MDS-UPDRS Part II Total Score
Description: For MDS-UPDRS Part II (motor experiences of daily living) scores, the scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 116
Units on a scale | 2.32 (0.335) | 0.13 (0.350)

4. Secondary Outcome: Change From Baseline in MDS-UPDRS Part III Total Score
Description: For MDS-UPDRS Part III (motor examination) scores, the scale range for Part III Total Score was 0-132, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 26 (LOCF)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 125 | 115
Units on a scale | -0.48 (0.639) | -4.47 (0.666)

5. Secondary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 117
Participants
  TEAEs | 66 | 73
  SAEs | 8 | 4

6. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs Values
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 117
Participants
  Temperature (<35.6 °C) | 20 | 17
  Temperature (>37.7 °C) | 1 | 0
  Systolic Blood Pressure (<90 mmHg) | 2 | 3
  Diastolic Blood Pressure (<50 mmHg) | 3 | 0
  Diastolic Blood Pressure (>100 mmHg) | 6 | 9
  Pulse (<45 bpm) | 0 | 1

7. Secondary Outcome: Number of Participants With TEAE Related to Body Weight
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 117
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With TEAE Related to Electrocardiograms (ECG)
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 117
Participants
  Extrasystoles | 0 | 1
  Myocardial infarction | 1 | 0
  Electrocardiogram QT prolonged | 0 | 1

9. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests
Time Frame: Up to Week 26
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TVP-1012 1mg
Number analyzed (Participants) | 126 | 117
Participants
  Blood creatine phosphokinase increased | 3 | 0
  Gamma-glutamyltransferase increased | 2 | 0
  Blood alkaline phosphatase increased | 1 | 0
  Glycosylated haemoglobin increased | 0 | 1
  Hepatic enzyme increased | 1 | 0
  Liver function test abnormal | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | TVP-1012 1mg
Serious Adverse Events (participants affected / at risk) | 8/126 | 4/117
Other Adverse Events (participants affected / at risk) | 24/126 | 23/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | TVP-1012 1mg (N=117)
Myocardial infarction (Cardiac disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=126) | TVP-1012 1mg (N=117)
Nasopharyngitis (Infections and infestations) | 19 | 18
Fall (Injury, poisoning and procedural complications) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.